CLINICAL TRIAL: NCT07117838
Title: Distractional Interventions on Patients' Anxiety, Pain and Physiological Parameters Durıng Coronary Angiography: The Effect of Virtual Reality and Music
Brief Title: Vırtual Reality and Music in Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HARUN ÜNAL (Other)
Responsible Party: Sponsor-Investigator, HARUN ÜNAL, Investigator, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1476
Record Dates: First submitted 2025-03-26; First posted 2025-08-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Virtual Reality; Nursing Caries
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: One count for 120 patients who met the study's inclusion criteria A list will be created and patients will be distributed to experimental and intervention groups with a computerized randomization program (https://www.random.org/integer-sets/). According to the randomization result, patients will be assigned to the virtual reality group (intervention 1), the music group (intervention 2) and the control group (Control) with standard treatment. All patients will be randomized to the intervention and control groups after being admitted to the angiography unit. - It will be named as intervention group (the group to which virtual reality glasses and music will be applied) and - Control group (the group to which no additional procedure will be applied to the standard care during the coronary angiography procedure).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality (Experimental): Patients were fitted with virtual reality glasses.
  Interventions: Other: virtual reality
- music (Experimental): Patients were listened to music
  Interventions: Other: music
- control (No Intervention): Patients were not interfered with and were receive standard care.

INTERVENTIONS:
Other: virtual reality — Virtual reality application were applied to patients during coronary angiography.
  Arms: virtual reality
Other: music — Patients will listen to music during coronary angiography.
  Arms: music

SUMMARY:
"Coronary The scope of this study, which was conducted for the purpose of "Distracting Interventions on Patients' Anxiety, Pain and Physiological Parameters During Angiography: The Effect of Virtual Reality and Music", is to help patients at the level of evidence during coronary angiography and to contribute to the literature.

DETAILED DESCRIPTION:
Before starting the application, patients who meet the criteria for inclusion in the study will be determined according to the randomization order and information about the study will be given.

Patients will be randomly assigned to the control and intervention groups (virtual reality and music group). Then, the following interventions will be applied sequentially, depending on the group the patient is included in.

After the appropriate participants are determined, written informed consent will be given to the participants and the Patient Introduction Form, State Anxiety Scale and Visual Comparison Scale will be applied just before the procedure begins, and then the patient's physiological parameters will be measured and recorded in the Patient Monitoring Form. Later patients will undergo coronary angiography. For the control group, conventional procedures will be applied by the researcher and medical care staff.

Patients in the virtual reality group, one of the intervention groups, will be shown a video with predetermined relaxing visuals and sounds through virtual reality glasses. Before watching the video, the researcher informed about the use of virtual reality glasses.

The patient will be informed. They will use the SG glasses for 3-5 minutes before the procedure begins for the patient to get used to it, and then the procedure will begin. VR glasses will be kept on throughout the procedure. In addition, the patient is advised at any stage of the application.

He will be told that he can remove his glasses and withdraw from the study. USB MP3 players and headphones will be provided by the researcher to collect data for the music group. Various styles of music (Classical World Music, Popular Music, Classical Turkish Music, Sufi Music) will be loaded into the USB MP3 player. Patients will be able to choose any of these music styles from the folder and listen to them. Music group patients from the intervention groups will be informed before starting the procedure and will be given 3-5 minutes.

MP3 reader and headphones will be provided throughout. Then, the patient will be taken to the coronary angiography procedure and will be allowed to listen to the previously prepared music of the patient's choice throughout the procedure.

Physiological parameters of patients during coronary angiography will be measured. After the procedure is completed, the Patient Introduction Form, State Anxiety Scale and Visual Comparison Scale will be applied to the patients in all three groups, and then the patient's physiological parameters will be measured and recorded in the Patient Monitoring Form.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 18-70, Patients who agreed to participate in the study voluntarily, Open to communication, Knows how to read and write, Patients without visual or auditory impairments, Patients who underwent femoral artery area intervention, Patients who are administered opioid and tranquilizer derivative drugs, Patients who were undergoing coronary angiography for the first time were included in the study.

Exclusion Criteria:

Having difficulty using virtual reality glasses, Patients with headache, nausea and vomiting were not included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | 10 minutes
  This form, prepared by researchers based on literature reviews, consists of a total of 13 questions to question the socio-demographic characteristics of patients and their disease-related characteristics.
Visual Analog Scale | 10 minutes
  The VAS, whose validity and reliability study was conducted by Price et al. (1983), is a tool that subjectively assesses and measures people's pain experiences. The VAS is frequently used in assessing pain levels in adults and is considered the fastest and simplest to understand among single-dimensional scales. To determine pain intensity, the patient is asked to mark the score corresponding to the quantitative pain experienced on a 10-cm ruler, with the "0" point at one end representing "no pain" and the "10" point at the other end representing "the most severe pain." The scale can be applied horizontally or vertically. The point marked by the patient is used as numerical data to determine the level of pain perception. On this scale, a "0" point indicates no pain, while a "10" point describes the most severe pain.
State Anxiety Scale | 10 minutes
  The study used the "State and Trait Anxiety Scale," developed by Spielberger et al. (1970) and translated and adapted into Turkish by Oner and Le Compte (1998). The scale consists of a total of 40 items and two separate scales. The first section includes the "State Anxiety Scale," which measures how a person feels in a given moment. The second section includes the "Trait Anxiety Scale," which also includes statements about how a person generally feels. This study was designed for use during coronary angiography, and the "State Anxiety Scale" was used based on literature research and expert opinions.
Patient Follow-up Form | 10 minutes
  This is a form created by researchers to record the physiological parameters (heart rate, respiratory rate, systolic blood pressure, diastolic blood pressure, oxygen saturation) measured by researchers before (manually), during (digitally via a femoral catheter), and after the procedure (digitally via a femoral catheter). The measurements taken from the patient were recorded on this form.

CONTACTS AND LOCATIONS:
Overall Officials: Harun ÜNAL, phd student, Study Chair — ataturk universty
Locations (1):
- Van Yuzuncu Yil University, Van, tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No